CLINICAL TRIAL: NCT00223418
Title: Do Patients Taking Aripiprazole Learn More in Vocational Skills Training Than Patients Taking Olanzapine?
Brief Title: Study Comparing Patients Taking Olanzapine and Patients Taking Aripiprazole on Learning of Vocational Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Dawn Velligan, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 023-0013-300
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Schizophenia Disorder; Schizoaffective Disorder
Keywords: aripiprazole; olanzapine; vocational; learning; cognition; cognitive
MeSH Terms: conditions — Psychotic Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
STUDY PURPOSE: To study whether patients who have schizophrenia or schizoaffective disorder and are randomly assigned to switch to aripiprazole prior to participation in a brief vocational skills training (VST) will have improved cognitive functioning and learn more in VST than those randomly assigned to stay on olanzapine. There is evidence that VST is important in improving role functioning for schizophrenia patients, however, cognitive impairments limit the ability of some patients to benefit from skills training approaches. Patients switched from olanzapine to aripiprazole improve in terms of verbal learning and verbal learning has been shown to be a strong predictor of community outcome. It is unclear whether the cognitive benefits of switching to aripiprazole extend to improve learning of vocational skills.

DETAILED DESCRIPTION:
Many schizophrenia outpatients have cognitive deficits and poor vocational functioning. There is evidence from randomized controlled trials that vocational skills training is important in improving vocational role functioning for schizophrenia patients. However, it has become clear that cognitive impairments limit the ability of patients to benefit from skills training approaches. Recent research demonstrates that patients switched from olanzapine to aripiprazole improve in terms of verbal learning. Verbal learning has been found to be a strong predictor of multiple domains of community outcome. It is unclear whether the cognitive benefits of switching to aripiprazole extend to improve learning of vocational skills. This study examines whether aripiprazole can improve the ability to benefit from expensive rehabilitation programs focused on skill-building. Specifically, the study examines whether patients who switch from olanzapine to aripiprazole learn more and benefit more from a brief vocational skills program than patients who remain on olanzapine. Specific aims are as follows: (1) we hypothesize that patients on aripiprazole will demonstrate better scores on tests of cognitive functioning following twelve weeks of medication treatment than patients on olanzapine and (2) we hypothesize that patients on aripiprazole will have significantly higher scores on vocational performance following a brief (2-day) vocational training and assessment session than those on olanzapine. Furthermore, we hypothesize that these gains will be maintained following one week of non-exposure to the trained vocational tasks.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Between ages of 18 and 52
* On olanzapine for a minimum of 3 months prior to participation
* Outpatient status for at least 3 months
* Vision and hearing intact or corrected to extent that will allow participation in vocational training and cognitive testing
* Score in impaired range on at least one test from a cognitive battery designed to be sensitive to impairments in schizophrenia
* Ability to participate in the informed consent process, as evidenced by an assessment of the capacity to give consent for research developed by the Maryland Psychiatric Research Center (DeRenzo et al., 1998).

Exclusion Criteria:

* History of head injury, mental retardation or neurological disorder
* Below a 4th grade reading level (32) according to the WRAT-3
* Taking multiple atypical antipsychotics
* Taking any decanoate antipsychotic
* Hospitalization in last 3 months
* Employment
* Alcohol or drug abuse that interferes with functioning or medication compliance

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2004-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Toilet Tank Assembly Task at 13 and 14 weeks
Card Sorting Task at baseline, 13 and 14 weeks

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale at baseline and 13 week
Negative Symptom Assessment at baseline and 13 week
Global Assessment of Functioning Scale at baseline and 13 week
Social and Occupational Functioning Scale at baseline and 13 week
Work portion of Test of Adaptive Behaviors in Schizophrenia at baseline and 13 week
STAN neurocognitive tests at baseline and 13 week
Trails A at baseline and 13 week
Trails Aa at baseline and 13 week
Trails B at baseline and 13 week

CONTACTS AND LOCATIONS:
Overall Officials: Dawn I Velligan, Ph.D., Principal Investigator — University of Texas Health Science Center in San Antonio; Mary D. Woolsey, M.S., Study Director — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States